CLINICAL TRIAL: NCT05048056
Title: A Phase 2, Multi-center, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy and Safety of AK120 in Adult Subjects With Moderate-to-Severe Atopic Dermatitis
Brief Title: Phase 2 Study of Efficacy and Safety of AK120, in Subjects With Moderate-to-Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical study and development strategy adjustment
Sponsor: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Akeso (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK120-203
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Monoclonal Antibodies
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AK120 Regimen 1 (Experimental): AK120 Regimen 1- subcutaneous injection every 2 weeks for 30 weeks.
  Interventions: Drug: AK120
- AK120 Regimen 2 (Experimental): AK120 Regimen 2- subcutaneous injection every 2 weeks for 30 weeks.
  Interventions: Drug: AK120
- Placebo to AK120 (Experimental): Placebo subcutaneous injection every 2 weeks, then crossover to AK120 Regimen 1, subcutaneous injection at Week16, after primary endpoint evaluation
  Interventions: Drug: Placebo; Drug: AK120

INTERVENTIONS:
Drug: Placebo — Placebo subcutaneous injection every 2 weeks for 16 weeks then Crossover to AK120 Regimen 1
  Arms: Placebo to AK120
Drug: AK120 — AK120 Regimen 1- subcutaneous injection every 2 weeks.
  Arms: AK120 Regimen 1; Placebo to AK120
Drug: AK120 — AK120 Regimen 2- subcutaneous injection every 2 weeks
  Arms: AK120 Regimen 2

SUMMARY:
This is a phase 2, multi-center, randomized, placebo-controlled, double-blind, parallel-group, dose-ranging study, conducted in subjects with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
This phase 2 study is designed to explore the efficacy and safety, as well as pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of dose-ranging AK120 compared to placebo, which will generate information regarding the selection of dosing regimens with AK120 monotherapy treatment in adult subjects with moderate-to-severe AD.

Primary Objectives:

• To evaluate the efficacy of AK120 in the treatment of adult subjects with moderate-to-severe Atopic Dermatitis (AD).

Secondary Objectives:

* To evaluate the safety of AK120 in the treatment of adult subjects with moderate-to-severe AD.
* To evaluate the Pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of AK120 in adult subjects with moderate-to-severe AD.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, over the age of 18
2. Chronic atopic dermatitis (AD) diagnosed at least 1 year.
3. Subject with EASI score ≥16, IGA ≥ 3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe), ≥ 10% body surface area (BSA) of AD involvement.
4. Subjects with a history of an inadequate response or medically inappropriate use of topical drug treatment within 6 months.

Key Exclusion Criteria:

1. Inadequate washout period for prior drug therapy (eg. corticosteroids, immunosuppressive/ immunomodulating, biologics, phototherapy, Chinese traditional medicine, anti-infective agents).
2. History of exposure to active TB, and/or history or current evidence of TB infection.
3. Positive serology results at Screening for hepatitis B, hepatitis C or HIV.
4. Any history of vernal keratoconjunctivitis (VKC) or atopic keratoconjunctivitis (AKC) within 6 months before the baseline visit.
5. History of clinical parasite infection, recent or planned travel to an area with endemic parasite infection within 6 months before the Screening visit
6. Any medical or psychiatric condition, laboratory, or ECG parameter which, in the opinion of the Investigator or the Sponsor's medical monitor, would place the subject at risk, interfere with participation in the study, or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving an Eczema Area and Severity Index (EASI) 75 response | At week 16

SECONDARY OUTCOMES:
Proportion of subjects achieving the Investigator Global Assessment (IGA, on a 5-point scale) for clear (0) or almost clear (1) | At week 16
Change in SCORing Atopic Dermatitis (SCORAD) | Baseline to Week 38
Change in Pruritus-Numerical Rating Scale (P-NRS) | Baseline to Week 38
Change in Body Surface Area (BSA) of AD involvement | Baseline to Week 38
Change in Patient Oriented Eczema Measure (POEM) | Baseline to Week 38
Individual subject AK120 concentrations in serum at different time points after AK120 administration | Baseline to Week 38
Change in pharmacodynamics studies TARC/CCL17 and IgE | Baseline to week 24
Anti-drug antibodies(ADAs) | Baseline to Week 38
Adverse events(AEs)/serious adverse events(SAEs) | Baseline to Week 38

CONTACTS AND LOCATIONS:
Locations (24):
- United States (16):
  - AkesoBio Investigative Site 2003, Little Rock, Arkansas
  - AkesoBio Investigative Site 2010, Canoga Park, California
  - AkesoBio Investigative Site 2021, San Diego, California
  - AkesoBio Investigative Site 2023, San Diego, California
  - AkesoBio Investigative Site 2017, San Francisco, California
  - AkesoBio Investigative Site 2020, Sherman Oaks, California
  - AkesoBio Investigative Site 2009, Hialeah, Florida
  - AkesoBio Investigative Site 2001, Hollywood, Florida
  - AkesoBio Investigative Site 2011, Miami, Florida
  - AkesoBio Investigative Site 2002, Weston, Florida
  - AkesoBio Investigative Site 2022, Ridgeland, Mississippi
  - AkesoBio Investigative Site 2015, Las Vegas, Nevada
  - AkesoBio Investigative Site 2013, Spartanburg, South Carolina
  - AkesoBio Investigative Site 2005, Rapid City, South Dakota
  - AkesoBio Investigative Site 2004, Houston, Texas
  - AkesoBio Investigative Site 2018, Houston, Texas
- Australia (3):
  - AkesoBio Investigative Site 3003, Sydney, New South Wales
  - AkesoBio Investigative Site 3002, Woolloongabba, Queensland
  - AkesoBio Investigative Site 3001, Camberwell, Victoria
- New Zealand (5):
  - AkesoBio Investigative Site 4003, Auckland
  - AkesoBio Investigative Site 4001, Auckland
  - AkesoBio Investigative Site 4005, Christchurch
  - AkesoBio Investigative Site 4004, Hamilton
  - AkesoBio Investigative Site 4004, Wellington

IPD SHARING:
Plan to Share IPD: No